CLINICAL TRIAL: NCT06135155
Title: A Single-center, Randomized, Double-blind, Parallel Design Phase Ⅰ Study to Compare the Pharmacokinetics of Two Different PEG-rhGH Preparations by Single Administration in Chinese Healthy Adult Male Subjects
Brief Title: A Clinical Trial to Compare Pharmacokinetics of Two Different PEG-rhGH Preparations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: GenSci004-102
Record Dates: First submitted 2023-10-31; First posted 2023-11-18 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2023-10

CONDITIONS: Pediatric Growth Hormone Deficiency (PGHD)
MeSH Terms: interventions — polyethylene glycol-recombinant human growth hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEG-rhGH with new preparation (Experimental)
  Interventions: Drug: PEG-rhGH with new preparation
- PEG-rhGH with present preparation (Experimental)
  Interventions: Drug: PEG-rhGH with present preparation

INTERVENTIONS:
Drug: PEG-rhGH with new preparation — A single subcutaneous injection of PEG-rhGH with new preparation
  Arms: PEG-rhGH with new preparation
Drug: PEG-rhGH with present preparation — A single subcutaneous injection of PEG-rhGH with present preparation
  Arms: PEG-rhGH with present preparation

SUMMARY:
The purpose of this study is to compare the pharmacokinetics of the two different PEG-rhGH preparations after a single administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male aged ≥18 years old and≤45 years old;
* The Body mass index (BMI): 19-26 kg/m2 (inclusive), and body weight ≥50 kg;
* Normal results of physical examination, vital signs, laboratory tests, 12 lead-ECG, chest X-ray, abdominal ultrasound, or non-clinical significance changes in the assessments above.

Exclusion Criteria:

* Subjects with a history of hypersensitivity reactions or clinically significant hypersensitivity reactions to drugs containing;
* Subjects with a clear history of disorders of the central nervous system, cardiovascular system, digestive system, respiratory system, urinary system, blood system, metabolic system, etc., or other diseases deemed unsuitable for participation in the trials by the investigators;
* Subjects with severe infection, severe trauma, or major surgery prior to screening;
* Subjects who have received blood transfusions, had blood donors, or lost blood before screening;
* Subjects who have positive results of human immunodeficiency virus antibodies (HIV-Ab), or hepatitis B surface antigen (HBsAg), or hepatitis C virus antibodies (HCV-Ab), or syphilis specific antibodies (TPPA);
* Subjects who have participated in clinical trials for medication or medical device prior to screening;etc.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2024-03-18 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (Peak Plasma Concentration (Cmax) ) of PEG-rhGH with present and new preparation | 0 hours -168 hours
Pharmacokinetics (Area under the concentration-time curve from time zero to time infinity (AUC0-∞)) of PEG-rhGH with present and new preparation | 0 hours -168 hours
Pharmacokinetics (Area under the concentration-time curve from time zero to time t (AUC0-t )) of PEG-rhGH with present and new preparation | 0 hours -168 hours

SECONDARY OUTCOMES:
Pharmacokinetics (The time to reach the peak drug concentration (Tmax)) of PEG-rhGH with present and new preparation. | 0 hours -168 hours
Pharmacokinetics (Half-life (t1/2)) of PEG-rhGH with present and new preparation. | 0 hours -168 hours
Pharmacokinetics (Terminal elimination rate constant (λz)) of PEG-rhGH with present and new preparation. | 0 hours -168 hours
Safety and tolerability（Number of participants with treatment-related adverse events） | 0 hours -168 hours
Safety and tolerability (Number of Participants with Abnormal Vital Signs That Are Related to Treatment) | 0 hours -168 hours
Safety and tolerability (Number of Participants with Abnormal 12-lead ECG QTc Interval That Are Related to Treatment) | 0 hours -168 hours
Safety and tolerability (Number of Participants with Abnormal Laboratory Values That Are Related to Treatment) | 0 hours -168 hours

OTHER OUTCOMES:
Anti-drug antibody (Number of Participants with positive ADA) | 0 hours -168 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Chengdu Xinhua Hospital affiliated to North Sichuan Medical College, Chengdu, Sichuan, China